CLINICAL TRIAL: NCT05893212
Title: Targeted Health Promotion With Guided Nature Walks or Group Exercise: a Controlled Trial in Primary Care
Brief Title: Nature Walks or Exercise as a Group Activity, the Effect Well-being, Sleep and Activity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Finnish Institute for Health and Welfare (Other Government); Municipality of Sipoo, Health and Social services (Unknown); Luonnontie (Unknown)
Responsible Party: Principal Investigator, Annika Kolster, Doctoral researcher, University of Helsinki
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUS/3520/2017
Record Dates: First submitted 2023-05-15; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Health Promotion; Multimorbidity
MeSH Terms: interventions — Exercise; Population Groups

STUDY DESIGN:
Intervention Model Description: This is a controlled pilot study on parallel groups in a real life, intention-to-treat setting.
Masking Description: Care provider recommended participation in either group, based on discussion with participant. All data is anonymized and stored at the Finnish Institute for Health and Welfare and outcomes assessor has access to this data, however, it includes knowledge of group participation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nature-group (Experimental): Primary care patients identified to be in the target group for health promoting activity by health or social service professionals. Participants chose to take part in the 8 week nature-group, meeting weekly in outdoor areas.
  Interventions: Behavioral: Nature based facilitated group intervention
- Sports-group (Active Comparator): Primary care patients identified to be in the target group for health promoting activity by health or social service professionals. Participants chose to take part in the 8 week sports-group, meeting weekly in community sports facilities.
  Interventions: Behavioral: Exercise in group

INTERVENTIONS:
Behavioral: Nature based facilitated group intervention — The Nature-group programme included learning more about local outdoor areas and nature itself, the biotopes visited were chosen to provide a various nature experience, including forests, farmland, lakes, and seashore. Accompanied by nature guides the group practiced simple sensorial exercises that enhance the contact with nature and its microbiome.
  Arms: Nature-group
Behavioral: Exercise in group — The Sports-group participated in an exercise programme and met weekly in community sports facilities. Exercise we define as a planned, structured, repetitive, and purposeful form of physical activity that aims for improvement or maintenance of one or more components of physical fitness. The sports programme was planned and executed by professional sports leaders in cooperation with health professionals and included both aerobic and anaerobic exercise as well as team sports, content was planned according to current best practice and considered the participants physical ability.
  Arms: Sports-group

SUMMARY:
Contact with nature promotes human wellbeing through diverse pathways, providing a potential way to support health especially in primary care, where patients commonly suffer from multimorbidity and poor general health. Social prescribing as a non-pharmaceutical treatment is a promising method to improve health as well as inclusion. This study explores and compares the effects of a nature based and an exercise based social prescribing scheme on mental wellbeing, physical activity and sleep, in a primary care population.

DETAILED DESCRIPTION:
In this non-randomized, intention-to-treat, pilot study we recruited clients at the health and social service centre in Sipoo, Finland.

Participants (n=79) chose between two social prescribing programs, either taking part of guided walks in nature, including immersion in a forest with high biodiversity, or taking part in a sports group with a versatile program. Inclusion was not based on diagnosis, but an identified need of improving health. Mental wellbeing was assessed using the 14-item Warwick-Edinburgh Mental Well-Being Scale (WEMWBS), additional questions evaluated perceived health and sleep. Amount and quality of sleep and physical activity were measured using wrist-worn accelerometers.

Assessments took place before and after the 8-week intervention, as we were interested in the effect on everyday life. Even though participants lived in an area with abundant green space, taking part in the prescribed nature program improved mental wellbeing. Those who initially rated their health and mental health as good did achieve benefit from both programs, while those in poor health received better aid from the nature group.

Initial study plan aimed for 160 participants, with an equal distribution between the groups. The programs were completed in 2018-2019 (spring + autumn) The COVID-19 outbreak hindered group activities 2020, a nature-group was organized in autumn 2020.

ELIGIBILITY:
Inclusion Criteria:

* Need of health promotion or secondary prevention of disease as identified by health care professionals or by social care professionals working in a public health care center (nurse, doctor, or social worker).
* Enrolment was not based on a diagnosis, but health care and social care professionals were instructed to identify patients/clients they felt could benefit from a targeted health intervention and involve particularly those in poor general health.
* Adults with a physical ability to slowly walk approximately 3 km in a slow tempo.
* Ability to understand and give consent to participation.
* Age 18 years or older.

Exclusion Criteria:

* Untreated medical condition hindering physical activity or symptomatic condition demanding continuous attention.
* Disability preventing ability to move in terrain.
* Inability to take part in group-based activities due to, e.g., behavioral challenges.

Although reason of referral is not reported, enrolment in intervention was part of real-life treatment.

Eligibility was assessed by professionals referring to the intervention, as well as at the introductory meeting organized by the staff at the public health care center taking place before the intervention started.

It was possible to take part in the intervention but not the study, participants in the study signed an informed consent allowing use of data and giving permission for later contact. Participants were free to withdraw from the study at any time without giving a reason, and this did not interfere with their care in any way.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in positive mental well-being | At beginning of study (day 0), 4.th meeting (day 28) and at end of study (day 56-58)
  Self-assessed mental wellbeing measured with the 14-item Warwick-Edinburgh Mental Well-Being Scale (WEMWBS).
Change in self rated health | At beginning of study (day 0), 4.th meeting (day 28) and at end of study (day 56-58)
  Question: How is your health at the moment? Likert-like scale: 1-5
Change in self rated mental health | At beginning of study (day 0), 4.th meeting (day 28) and at end of study (day 56-58)
  Question: How is your mental health at the moment? Likert-like scale: 1- 5 (much/good/well).
Change in functioning ability | At beginning of study (day 0), 4.th meeting (day 28) and at end of study (day 56-58)
  Question: How is your functioning ability at the moment? Likert-like scale: 1-5
Change in percieved sleep | At beginning of study (day 0), 4.th meeting (day 28) and at end of study (day 56-58)
  Question: How do you sleep at the moment? Likert-like scale: 1-5

SECONDARY OUTCOMES:
Change in total sleep time | Before starting intervention (day 0) and after intervention (day 56-60)
  For objective measurement of amount and quality of activity and sleep, participants kept a wrist worn accelerometer (ActiGraph GT9X Link, Actigraph LLC, Pensacola, Florida, USA).
  Sleep is reported total sleep time, time in bed and sleep efficiency. After sleep onset the number and length of awakenings is also reported.
Change in time in bed. | Before starting intervention (day 0) and after intervention (day 56-60)
  For objective measurement of amount and quality of activity and sleep, participants kept a wrist worn accelerometer (ActiGraph GT9X Link, Actigraph LLC, Pensacola, Florida, USA).
  Sleep is reported total sleep time, time in bed and sleep efficiency. After sleep onset the number and length of awakenings is also reported.
Change in sleep efficiency | Before starting intervention (day 0) and after intervention (day 56-60)
  For objective measurement of amount and quality of activity and sleep, participants kept a wrist worn accelerometer (ActiGraph GT9X Link, Actigraph LLC, Pensacola, Florida, USA).
  Sleep is reported total sleep time, time in bed and sleep efficiency. After sleep onset the number and length of awakenings is also reported.
Change in number and length of awakenings after sleep onset | Before starting intervention (day 0) and after intervention (day 56-60)
  For objective measurement of amount and quality of activity and sleep, participants kept a wrist worn accelerometer (ActiGraph GT9X Link, Actigraph LLC, Pensacola, Florida, USA).
  After sleep onset the number and length of awakenings is also reported.
Change in light physical activity | Before starting intervention (day 0) and after intervention (day 56-60)
  For objective measurement of amount and quality of activity and sleep, participants kept a wrist worn accelerometer (ActiGraph GT9X Link, Actigraph LLC, Pensacola, Florida, USA). As we are interested in the effects on everyday life, accelerometer data was not collected during the intervention itself, but before starting the program and after the intervention. Data shows the number of active days with the minimum of 10 hours of wear time from midnight-to-midnight, where the activity levels are divided in light (LPA), moderate (MPA) and vigorous (VPA) intensity.
  Accelerometers of the same type have been used in the population-based health examination study FinHealth 2017 Survey, providing us with a meaningful reference when interpreting the data.
Change in moderate physical activity | Before starting intervention (day 0) and after intervention (day 56-60)
  For objective measurement of amount and quality of activity and sleep, participants kept a wrist worn accelerometer (ActiGraph GT9X Link, Actigraph LLC, Pensacola, Florida, USA). As we are interested in the effects on everyday life, accelerometer data was not collected during the intervention itself, but before starting the program and after the intervention. Data shows the number of active days with the minimum of 10 hours of wear time from midnight-to-midnight, where the activity levels are divided in light (LPA), moderate (MPA) and vigorous (VPA) intensity.
  Accelerometers of the same type have been used in the population-based health examination study FinHealth 2017 Survey, providing us with a meaningful reference when interpreting the data.
Change in vigorous physical activity | Before starting intervention (day 0) and after intervention (day 56-60)
  For objective measurement of amount and quality of activity and sleep, participants kept a wrist worn accelerometer (ActiGraph GT9X Link, Actigraph LLC, Pensacola, Florida, USA). As we are interested in the effects on everyday life, accelerometer data was not collected during the intervention itself, but before starting the program and after the intervention. Data shows the number of active days with the minimum of 10 hours of wear time from midnight-to-midnight, where the activity levels are divided in light (LPA), moderate (MPA) and vigorous (VPA) intensity.
  Accelerometers of the same type have been used in the population-based health examination study FinHealth 2017 Survey, providing us with a meaningful reference when interpreting the data.
Change in importance of nature and physical activity | Before starting intervention (day 0) and after intervention (day 56)
  Question: Is nature important to you? Likert-like scale:1-5
Change in importance physical activity | Before starting intervention (day 0) and after intervention (day 56)
  Question: Is physical exercise important to you? Likert-like scale: 1- 5

CONTACTS AND LOCATIONS:
Overall Officials: Timo Partonen, MD, PhD, Study Director — Research professor at Finnish Institute for Health and Welfare
Locations (1):
- Sipoo Social and Health center, Sipoo, Itä-Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No
According to the original research permission granted by the Finnish Institute for Health and Welfare all data is anonymized and stored at the institute, only accessible to researchers with permission from the institute.

REFERENCES:
- [Derived] Kolster A, Heikkinen M, Pajunen A, Mickos A, Wennman H, Partonen T. Targeted health promotion with guided nature walks or group exercise: a controlled trial in primary care. Front Public Health. 2023 Aug 24;11:1208858. doi: 10.3389/fpubh.2023.1208858. eCollection 2023. PMID 37766747
- See also: Master's thesis, Heikkinen, Malin (2022) Hälsofrämjande Hälsoskog gruppverksamhet i Sibbo kommuns social- och hälsovårdstjänster: upplevelser ur ett deltagarperspektiv — https://urn.fi/URN:NBN:fi:amk-2022121429968